CLINICAL TRIAL: NCT07108829
Title: First-in-Man Clinical Study to Evaluate the Safety and Efficacy of Renal Artery Radiofrequency Ablation Clamp, Radiofrequency Ablation Generator for the Adjunctive Treatment of Refractory Hypertension and Drug-Intolerant Hypertension
Brief Title: Laparoscopic Adventitial Renal Denervation (RDN) for Refractory Hypertension
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Henan Institute of Cardiovascular Epidemiology (Other)
Collaborators: Hunan Ept Medical Co., Ltd. (Unknown); Shanghai Hongtong Industrial Co., Ltd. (Unknown)
Responsible Party: Principal Investigator, Chuanyu Gao, Professor, Henan Institute of Cardiovascular Epidemiology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HenanlCE202503
Record Dates: First submitted 2025-07-31; First posted 2025-08-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-07

CONDITIONS: Refractory Hypertension or Drug-intolerant Hypertension
Keywords: Hypertension; Resistant Hypertension; Renal Denervation; Laparoscopic; Radiofrequency Ablation; Sympathetic Nerves
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Laparoscopic Adventitial RDN (Experimental): Participants will undergo a 28-day run-in period on a standardized antihypertensive medication regimen. Following this period, all participants will receive the investigational treatment, which is a laparoscopic renal artery adventitial denervation procedure. Participants will be followed for 180 days post-procedure
  Interventions: Device: Renal Artery Radiofrequency Ablation Clamp

INTERVENTIONS:
Device: Renal Artery Radiofrequency Ablation Clamp — This device is a clamp used during a laparoscopic surgical procedure. It is placed on the external surface (adventitia) of the renal artery and is connected to a radiofrequency generator. It delivers targeted radiofrequency energy to ablate the renal sympathetic nerves.

SUMMARY:
This is a first-in-human study to test the safety and effectiveness of a new device-based treatment for high blood pressure that is difficult to control with medicine. This condition is known as refractory hypertension.

The study will enroll 10 adults aged 18 to 65 whose high blood pressure is not controlled even though they are taking three or more blood pressure medications.

The treatment involves a new medical device called a Renal Artery Radiofrequency Ablation Clamp. This device is used during a keyhole (laparoscopic) surgery. It works by applying controlled heat (radiofrequency energy) to the outside of the arteries that supply blood to the kidneys. This procedure, known as renal denervation, aims to calm the nerves around these arteries that contribute to high blood pressure.

Participants who join the study will first be monitored on a standard set of blood pressure medicines to confirm they are eligible. If they qualify, they will undergo the keyhole surgery. After the procedure, participants will be followed for 180 days (about 6 months) and will have several follow-up visits to check their blood pressure and overall health.

DETAILED DESCRIPTION:
Rationale: Hypertension is a leading risk factor for cardiovascular disease. A significant portion of patients have refractory hypertension, where blood pressure remains elevated despite the use of multiple antihypertensive medications. The renal sympathetic nervous system plays a crucial role in blood pressure regulation, and its overactivity is a key factor in hypertension. Renal Denervation (RDN) is a device-based therapy designed to lower blood pressure by ablating these nerves. While most existing RDN systems use an endovascular (inside the artery) approach, this method carries potential risks such as endothelial damage, thrombosis, or renal artery stenosis.

Study Objective and Design: This is a prospective, single-center, single-arm, first-in-man (FIM) clinical study designed to provide a preliminary evaluation of the safety and efficacy of a novel laparoscopic adventitial RDN system for treating refractory or drug-intolerant hypertension. A total of 10 subjects will be enrolled. The study aims to gather initial feasibility and safety data to support the design of future, larger clinical trials.

Intervention: The investigational procedure is a laparoscopic renal artery adventitial RDN. This technique involves placing a Renal Artery Radiofrequency Ablation Clamp around the external surface (adventitia) of the main renal arteries. A compatible radiofrequency generator delivers energy to the clamp's electrodes, creating targeted lesions to ablate the sympathetic nerves while preserving the integrity of the arterial wall.

Methodology: Potential subjects will be screened for eligibility. Qualified candidates will enter a 28-day run-in period where they will be treated with a standardized, fixed-dose combination of at least three antihypertensive drugs, including a diuretic. This period is to confirm refractory status and assess medication adherence, which is confirmed via urine analysis. Subjects who still meet the blood pressure criteria after the run-in period will undergo the laparoscopic RDN procedure. Post-procedure, subjects will be followed at discharge (or Day 7), Day 30, Day 90, and Day 180. Antihypertensive medications may be adjusted after 90 days according to a predefined protocol based on blood pressure response. Efficacy will be assessed by changes in office and 24-hour ambulatory blood pressure, as well as changes in medication burden. Safety will be monitored by tracking the incidence of Major Adverse Events (MAE), procedure-related complications, and changes in renal function throughout the 180-day follow-up period.

ELIGIBILITY:
Inclusion Criteria:

Age ≥18 years and ≤65 years, any sex.

Diagnosed with primary hypertension.

History of hypertension for at least 6 months.

Blood pressure meets the following two conditions:

Office systolic blood pressure ≥140mmHg and ≤180mmHg, and office diastolic blood pressure ≥90mmHg. If not taking a beta-blocker, resting heart rate must be ≥70bpm.

24-hour ambulatory blood pressure measurement shows an average systolic pressure ≥130mmHg or a daytime average systolic pressure ≥135mmHg.

Has a history of antihypertensive medication use within the last 6 months with uncontrolled blood pressure. Before enrollment, must undergo at least 28 days of a standardized medication regimen (including a diuretic and at least three drugs in total) with ≥80% compliance, while office SBP remains ≥140mmHg and ≤180mmHg, and office DBP remains ≥90mmHg.

Patient is willing and able to comply with follow-up requirements and has signed the informed consent form.

Exclusion Criteria:

Secondary hypertension.

Target renal artery anatomy is unsuitable, including:

Renal artery diameter >9mm or <4mm.

Multiple renal arteries.

Severe calcification, stenosis >50%, malformation, fibromuscular dysplasia, or aneurysm in either renal artery.

History of renal artery intervention (e.g., balloon angioplasty or stenting).

Unsuitable for laparoscopic surgery via the retroperitoneal approach, including prior retroperitoneal surgery, retroperitoneal fibrosis, or severe obesity (BMI > 40 kg/m²).

History of kidney transplant or severe renal impairment (eGFR < 45 mL/min/1.73m²).

Hospitalization for a hypertensive crisis within the past year.

Severe liver dysfunction (ALT or AST > 3 times the upper limit of normal).

Type 1 diabetes.

History of a cardiovascular event (e.g., myocardial infarction, unstable angina) or cerebrovascular event (e.g., stroke, TIA) within the last 6 months.

Pregnancy or planning to become pregnant during the trial.

Participation in any other investigational drug or device trial within 3 months prior to screening.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Rate of Achieving Target Office Systolic Blood Pressure at 180 Days | 180 days post-procedure
  The percentage of subjects whose office systolic blood pressure (SBP) is less than 140mmHg at the 180-day post-procedure follow-up. Office blood pressure will be measured in a resting state according to a standardized procedure.
Change From Baseline in Antihypertensive Medication Composite Score at 180 Days | 180 days post-procedure
  The change from baseline in a composite score reflecting the type and dose of antihypertensive medication required to achieve a target office SBP of <140mmHg. The score is calculated as (number of drug classes) multiplied by (the sum of the doses), where a standard daily dose is defined as 1, a half dose is 0.5, and a double dose is 2. The change is calculated as the baseline score minus the 180-day score.

SECONDARY OUTCOMES:
Procedural Success Rate | Intra-procedural
  The percentage of procedures where the renal artery radiofrequency ablation clamp is successfully positioned and the denervation procedure is completed without related complications, which include renal artery perforation and renal artery embolism.
Change From Baseline in Mean 24-hour Ambulatory Systolic Blood Pressure at 180 Days | Baseline and 180 days post-procedure
  The reduction in mean 24-hour ambulatory systolic blood pressure (SBP) at 180 days post-procedure compared to the baseline measurement.
Incidence of Major Adverse Events (MAE) | Up to 180 days post-procedure
  The percentage of subjects experiencing one or more Major Adverse Events. MAEs include all-cause mortality, new myocardial infarction, major bleeding, end-stage renal disease, major embolic events causing end-organ damage, renal artery re-intervention, renal artery perforation or dissection, vascular complications requiring intervention, hospitalization for hypertensive crisis, new stroke, or new-onset renal artery stenosis (≥70%).
Incidence of Laparoscopic Surgery-Related Adverse Events | Up to 30 days post-procedure
  The percentage of subjects experiencing adverse events related to the laparoscopic procedure. These include pneumoperitoneum-related complications (e.g., gas embolism, pneumothorax), injury to major abdominal or retroperitoneal vessels, visceral injury (bowel, bladder, liver, spleen), or ureteral injury.

CONTACTS AND LOCATIONS:
Locations (1):
- Fuwai Huazhong Cardiovascular Hospital, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No
The protocol's confidentiality section states that all study content and data are confidential and the exclusive property of the sponsor. It specifies that this information cannot be disclosed to any third party without the sponsor's consent , and this obligation of confidentiality remains in effect even after the trial is completed. This indicates there is no plan to share individual participant data.

REFERENCES:
- [Background] Gao C, Zhao L, Zhu L, Li M, Ding D, Liu Z, Fan Z, Zhang Y, Zhao W, Wang J. Laparoscopic-based perivascular unilateral renal sympathetic nerve denervation for treating resistant hypertension: a case report. Hypertens Res. 2019 Aug;42(8):1162-1165. doi: 10.1038/s41440-019-0237-3. Epub 2019 Feb 27. PMID 30814662
- [Background] Baik J, Song WH, Yim D, Lee S, Yang S, Lee HY, Choi EK, Jeong CW, Park SM. Laparoscopic Renal Denervation System for Treating Resistant Hypertension: Overcoming Limitations of Catheter-Based Approaches. IEEE Trans Biomed Eng. 2020 Dec;67(12):3425-3437. doi: 10.1109/TBME.2020.2987531. Epub 2020 Nov 19. PMID 32310758
- [Background] Liu Y, Zhu B, Zhu L, Zhao L, Ding D, Liu Z, Fan Z, Zhao Q, Zhang Y, Wang J, Gao C. Clinical outcomes of laparoscopic-based renal denervation plus adrenalectomy vs adrenalectomy alone for treating resistant hypertension caused by unilateral aldosterone-producing adenoma. J Clin Hypertens (Greenwich). 2020 Sep;22(9):1606-1615. doi: 10.1111/jch.13963. Epub 2020 Aug 18. PMID 32812324
- [Background] Zhao L, Su E, Yang X, Zhu B, Fan Z, Wang X, Qi D, Zhu L, Bai M, Zhang Y, Zhao Q, Li M, Gao C. Laparoscopic-based perivascular renal sympathetic nerve denervation: a feasibility study in a porcine model. Eur J Med Res. 2020 Jun 18;25(1):22. doi: 10.1186/s40001-020-00422-5. PMID 32552871
- [Background] Krum H, Schlaich M, Whitbourn R, Sobotka PA, Sadowski J, Bartus K, Kapelak B, Walton A, Sievert H, Thambar S, Abraham WT, Esler M. Catheter-based renal sympathetic denervation for resistant hypertension: a multicentre safety and proof-of-principle cohort study. Lancet. 2009 Apr 11;373(9671):1275-81. doi: 10.1016/S0140-6736(09)60566-3. Epub 2009 Mar 28. PMID 19332353